CLINICAL TRIAL: NCT07346599
Title: The Effect of Bilateral Lumbar Erector Spinae Plane Block on Postoperative Analgesia in Lumbar Spinal Surgery
Brief Title: A Block Method for Pain After Back Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya City Hospital (Other)
Responsible Party: Principal Investigator, MERVE KAYNAK, specialist doctor, Afyonkarahisar Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 448
Record Dates: First submitted 2025-12-09; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Nerve Block; Postoperative Pain; Randomised Clinical Trial
Keywords: POSTOPERATİVE PAİN; ERECTOR SPİNA PLANE BLOCK; LUMBAR SPİNAL SURGERY
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESP BLOCK, (Active Comparator)
  Interventions: Procedure: ESP block group
- CONTROL GROUP (No Intervention)

INTERVENTIONS:
Procedure: ESP block group — BILATERAL TWO-LEVEL ESP BLOCK WAS APPLIED TO PATIENTS UNDERGOING LUMBAR SPINAL SURGERY.
  Arms: ESP BLOCK,

SUMMARY:
The purpose of this clinical trial is to evaluate whether bilateral lumbar erector spinae plane (ESP) block can reduce postoperative pain in adult patients undergoing lumbar spine surgery. The study also assesses the safety of this method and its effects on the recovery process. The main questions it aims to answer are:

Do patients who receive the ESP block experience less postoperative pain? Do these patients require fewer opioid (morphine-derived) analgesics? Does the first analgesic requirement occur later? Do patients mobilize earlier (stand/walk sooner)? Does the ESP block affect hemodynamic stability during and after surgery? Researchers will compare the ESP block group with the standard analgesia group to determine whether these effects occur.

Participants:

Patients in this study will be asked to:

Be randomly assigned to one of two groups before lumbar spine surgery Receive either a bilateral ESP block or standard analgesic therapy

Undergo postoperative follow-up including:

measurement of pain scores, recording of analgesic consumption, assessment of time to first analgesic requirement, monitoring of mobilization time, valuation of possible side effects

DETAILED DESCRIPTION:
This randomized controlled study was designed to evaluate the effect of bilateral lumbar erector spinae plane (ESP) block on postoperative analgesia in patients undergoing lumbar spine surgery. A total of 102 patients scheduled for lumbar spine surgery were enrolled in the study and randomly assigned into two groups. One group received a bilateral ESP block at the L2-L4 levels using 20 mL of 0.25% bupivacaine on each side, while the control group received standard postoperative analgesia.

Postoperative pain assessment, opioid consumption, time to first analgesic request, mobilization time, intraoperative hemodynamic parameters, and the occurrence of adverse events were prospectively recorded according to a predefined follow-up protocol. The study was conducted using a prospective, randomized design to assess the efficacy and safety of bilateral lumbar ESP block for postoperative pain management in lumbar spine surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and over, 80 and under
* American Society of Anesthesiologists Patient Classification Score (ASA) between I and Ⅲ
* Patients who can cooperate and give consent
* No chronic analgesic or opioid use
* No mental or psychiatric disorders
* No alcohol or illicit drug use
* Patients scheduled for elective spinal surgery

Exclusion Criteria:

* -Patients who withdrew from participation at any time during the study
* Foreign nationals who could not be contacted
* Patients under 18 and over 80
* Patients with an ASA score of Ⅳ or higher
* Patients scheduled for emergency surgery
* Pregnant women and breastfeeding mothers
* Bleeding diathesis
* Drug allergy
* Anticoagulant use
* Local/systemic infection
* Serious arrhythmia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
VAS values of patients in the first 24 hours postoperatively | The first 24 hours postoperatively
  Zero indicates no pain, and 10 indicates the worst possible pain

CONTACTS AND LOCATIONS:
Overall Officials: merve kaynak, Principal Investigator — Kütahya City Hospital; Ali Kaynak, Study Chair — Kütahya City Hospital; bilal a bezen, Study Chair — Afyonkarahisar Health Sciences University Hospital; remziye sıvacı, Study Director — Afyonkarahisar Health Sciences University Hospital; elif d bakı, Study Chair — Afyonkarahisar Health Sciences University Hospital; serhat yıldızhan, Study Chair — Afyonkarahisar Health Sciences University Hospital
Locations (1):
- Afyonkarahisar Health Sciences University Hospital, Afyonkarahisar, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Result] Goel VK, Chandramohan M, Murugan C, Shetty AP, Subramanian B, Kanna RM, Rajasekaran S. Clinical efficacy of ultrasound guided bilateral erector spinae block for single-level lumbar fusion surgery: a prospective, randomized, case-control study. Spine J. 2021 Nov;21(11):1873-1880. doi: 10.1016/j.spinee.2021.06.015. Epub 2021 Jun 23. PMID 34171466
- [Result] Tseng V, Xu JL. Erector Spinae Plane Block for Postoperative Analgesia in Lumbar Spine Surgery: Is There a Better Option? J Neurosurg Anesthesiol. 2021 Jan;33(1):92. doi: 10.1097/ANA.0000000000000631. No abstract available. PMID 31343504
- [Result] Liu H, Zhu J, Wen J, Fu Q. Ultrasound-guided erector spinae plane block for postoperative short-term outcomes in lumbar spine surgery: A meta-analysis and systematic review. Medicine (Baltimore). 2023 Feb 17;102(7):e32981. doi: 10.1097/MD.0000000000032981. PMID 36800574

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-24): https://cdn.clinicaltrials.gov/large-docs/99/NCT07346599/Prot_SAP_000.pdf
  • Informed Consent Form (2021-08-24): https://cdn.clinicaltrials.gov/large-docs/99/NCT07346599/ICF_001.pdf